CLINICAL TRIAL: NCT04222699
Title: Cultures Before and After Decolonization in Community Dwelling Adults With Current S. Aureus Colonization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: INFB-018-01CX
Record Dates: First submitted 2019-12-23; First posted 2020-01-10 (Actual); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Human Microbiome
Keywords: intranasal mupirocin; topical chlorhexidine
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intranasal Mupirocin and Topical Chlorhexidine (Experimental): Antimicrobial antiseptic skin cleanser (4% chlorhexidine) for daily use on Day 1, 3 and 5 of Week 8 of the study. BACTROBAN NASAL ointment (mupirocin calcium ointment, 2%) for use intranasally twice-daily on Day 1, 2, 3, 4 and 5 of Week 8 of the study.
  Interventions: Drug: Mupirocin calcium ointment, 2%; Drug: Topical Chlorhexidine, 4%

INTERVENTIONS:
Drug: Mupirocin calcium ointment, 2% — Mupirocin nasal ointment is used to treat or prevent infections in the nose due to certain strains of Staphylococcus aureus bacteria. This medicine works by killing bacteria or preventing their growth.
  Other Names: BACTROBAN NASAL ointment
Drug: Topical Chlorhexidine, 4% — Chlorhexidine is an antiseptic that fights bacteria.
  Topical chlorhexidine is used to clean the skin to prevent infection that may be caused by surgery, injection, or skin injury.

SUMMARY:
The investigators propose to study the microbiome of the nose, throat and three skin sites in a population without current exposure to the healthcare environment: 80 community dwelling adults. We will characterize the microbial communities in these body sites (nose, throat, perirectal and three skin sites) over time using culture-independent techniques. The investigators will then "decolonize" the subjects. Subjects will receive intranasal mupirocin and topical chlorhexidine. The investigators will then compare the microbial communities at baseline and after decolonization within individuals. Our overall hypothesis is that the microbial composition of these sites and the response to decolonization is influenced by the healthcare environment and that decolonization leads to re-colonization with an increasing proportion of Gram-negative bacilli.

ELIGIBILITY:
Inclusion Criteria:

* Veteran living in the greater Baltimore, MD area
* Adults >= 18 years of age
* Living independently
* Willing and able to provide anterior nares, skin, throat, and perirectal specimens over an 18 week time period.
* Willing and able to administer intranasal mupirocin and topical chlorhexidine over a five day period
* Capable of understanding and complying with the entire study protocol.
* Provided signed and dated informed consent

Exclusion Criteria:

* Use of anticancer chemotherapy or radiation therapy (cytotoxic) within the past 6 months
* History of HIV infection with most recent CD4 of <200
* Immunosuppression medications within the past 3 months
* Use of systemic antibacterial or antifungal agents in the past 3 months
* Use of nasal steroids currently or in the past 3 months
* Use of nasal antimicrobial ointment in the past 3 months
* Any current indwelling percutaneous medical device or urinary catheter
* Acute care hospitalization in the past 3 months
* Planned surgery or hospitalization during the study period
* History of an allergic reaction to chlorhexidine or mupirocin
* Oral temperature of >100 F at enrollment visit
* BMI <18 or >35 at enrollment visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-09-18 (Actual); Primary Completion 2014-11-18 (Actual); Study Completion 2014-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Claire Roghmann, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants were S. aureus negative in the nose at enrollment and were withdrawn from the study as the use of mupirocin was not clinically indicated.
Groups:
- Intranasal Mupirocin and Topical Chlorhexidine: Antimicrobial antiseptic skin cleanser (4% chlorhexidine) for daily use on Day 1, 3 and 5 of Week 8 of the study. BACTROBAN NASAL ointment (mupirocin calcium ointment, 2%) for use intranasally twice-daily on Day 1, 2, 3, 4 and 5 of Week 8 of the study.
  Mupirocin calcium ointment, 2%: Mupirocin nasal ointment is used to treat or prevent infections in the nose due to certain strains of Staphylococcus aureus bacteria. This medicine works by killing bacteria or preventing their growth.
  Topical Chlorhexidine, 4%: Chlorhexidine is an antiseptic that fights bacteria.
  Topical chlorhexidine is used to clean the skin to prevent infection that may be caused by surgery, injection, or skin injury.
Period: Overall Study
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Started | 28
Completed | 26
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in the Abundance of Staphylococcus Aureus in the Nose After Decolonization
Description: Change in the abundance of Staphylococcus aureus in the nose from immediately before mupirocin administration to 8 weeks after mupirocin administration.
Time Frame: 8 weeks
Population: Out of the 28 participants assigned to this group, 2 were lost to follow-up and 1 had an insufficient amount of sample collected and could not be included in the analysis.
Measure: Mean (Standard Deviation); unit: fg/uL
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 25
fg/uL | -781 (3681)

2. Primary Outcome: Change in the Abundance of Staphylococcus Aureus in the Throat After Decolonization
Description: Change in the abundance of Staphylococcus aureus in the throat from immediately before mupirocin administration to 8 weeks after mupirocin administration.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fg/uL
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 25
fg/uL | -321 (7053)

3. Primary Outcome: Change in the Abundance of Gram Negative Bacteria on the Subclavian Skin After Decolonization
Description: Quantitative PCR using 16S rRNA is used to quantify the total bacterial load of Gram negative bacteria on the subclavian skin before and after decolonization.
Time Frame: 12 months
Population: Subclavian skin samples deteriorated prior to sample analysis and cannot be used.
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 0

4. Primary Outcome: Change in the Abundance of Gram Negative Bacteria on the Femoral Skin After Decolonization
Description: Quantitative PCR using 16S rRNA is used to quantify the total bacterial load of Gram negative bacteria on the femoral skin before and after decolonization.
Time Frame: 12 months
Population: Femoral skin samples deteriorated prior to sample analysis and cannot be used.
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes